CLINICAL TRIAL: NCT01026441
Title: Clinical Study to Evaluate the Safety and Efficacy of the Vela100/eShape Uno Device for Cellulite and Circumference Reduction
Brief Title: Clinical Study to Evaluate the Safety and Efficacy of the Vela100
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Product was not developed and study was cancelled
Sponsor: Syneron Medical (Industry)
Responsible Party: VP Research and Development, Syneron
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vela100
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Cellulite Reduction; Circumference Reduction
Keywords: Aesthetic

ARMS (1):
- Treatment for cellulite and circumference reduction (Other): All subjects will be treated with the device
  Interventions: Device: Vela100 (Aesthetic)

INTERVENTIONS:
Device: Vela100 (Aesthetic) — 6 treatments once a week

SUMMARY:
This study is intended to test the safety of the Vela100 device when used for treatment for cellulite and circumference temporary reduction.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent agreement signed by the subject.
* Healthy males or females older than 21 years of age but not older than 60 years of age.
* Fitzpatrick Skin Type I to VI
* Having at least two areas (abdomen, buttocks and thighs) suitable for treatment.
* BMI score is greater than 18.5 and less than 29.9 - normal to overweight, but not obese.
* Willingness to follow the treatment and follow-up schedule and the post-treatment care.
* Willingness to refrain from a change in diet/drinking/exercise/medication regimen for the entire course of the study.
* For female of child bearing potential - using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study (i.e., oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide, or abstinence).

Exclusion Criteria:

* Pregnant or planning to become pregnant, having given birth (vaginal birth or Caesarean surgery) less than 9 months ago, and/or breastfeeding.
* Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator.
* Having a permanent implant in the treated areas, such as metal plates and screws or an injected chemical substance.
* Having received treatment with laser, RF or other devices in the treated areas within 6 months of treatment or during the study.
* Having undergone a liposuction surgery or any contouring treatment in the areas intended for treatment within 9 months of treatment or during the study.
* For post-liposuction areas, the procedure should also not have been performed more than 2 years prior to this study.
* Having undergone any other surgery in the treated areas within 9 months of treatment or during the study.
* Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions.
* Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), lupus, porphyria, or pertinent neurological disorders.
* Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician discretion).
* History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
* Suffering from hormonal imbalance which may affect weight or cellulite, as per the Investigator's discretion.
* History of significant lymphatic drainage problems. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course.
* History of keloid scarring or of abnormal wound healing.
* History of being especially prone to bruising.
* History of epidermal or dermal disorders (particularly if involving collagen or microvascularity).
* Use of isotretinoin (Accutane®) within 6 months of treatment or during the study.
* Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) during, as well as two weeks before and after, the treatment course.
* Use of anti-cellulite creams within a month of treatment or during the course of the study.
* If any allergy that is related to the lotion used in this study appears, subjects may be excluded from the study.
* Recently tanned in areas to be treated and/or unable or unlikely to refrain from tanning during the study.
* Significant change in diet or exercise regimen within a month of enrollment or during this study and/or weight loss or gain of 10 lbs (4.5 kgs) within 2 months of enrollment or during this study.
* Participation in a study of another device or drug within 1 month prior to enrollment or during this study.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Adverse Events | End of treatment, at 1 month FU

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orange Coast Women's Medical Group, Laguna Hills, California
  - Kavali Plastic Surgery and Skin Renewal Center, Atlanta, Georgia